CLINICAL TRIAL: NCT01850108
Title: A Non-Myeloablative Conditioning and Transplantation of Partially HLA-Mismatched and HLA-Matched Bone Marrow for Patients With Sickle Cell Disease and Other Hemoglobinopathies
Brief Title: Non-Myeloablative Conditioning and Bone Marrow Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Responsible Party: Principal Investigator, Adetola A. Kassim, Professor of Medicine; Clinical Director, Sickle Cell Anemia Program; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICCNCCTT12108
Record Dates: First submitted 2013-05-01; First posted 2013-05-09 (Estimated); Results first posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Sickle Cell Disease; Hemoglobinopathies
MeSH Terms: conditions — Anemia, Sickle Cell; Hemoglobinopathies | interventions — thymoglobulin; fludarabine; fludarabine phosphate; Cyclophosphamide; Mesna; Sirolimus; Mycophenolic Acid; Bone Marrow Transplantation; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Non-Myeloablative Conditioning and Bone Marrow Transplantation (Experimental)
  Interventions: Drug: Thymoglobulin; Drug: Fludarabine; Drug: Cyclophosphamide (CTX); Drug: Mesna; Drug: Sirolimus; Drug: Mycophenolate mofetil (MMF); Procedure: Bone marrow transplantation; Radiation: Total body irradiation

INTERVENTIONS:
Drug: Thymoglobulin — Day 9 before BMT: 0.5mg/kg IV; Days 8 & 7 before BMT: 2mg/kg IV
  Days 8 & 7 - 2mg/kg IV before BMT
Drug: Fludarabine — Days 6 and 2 before BMT: 30mg/m2/day IV
  Other Names: Fludara®
Drug: Cyclophosphamide (CTX) — Days 6 and 5 before BMT: 14.5mg/kg IV; Days 3 and 4 after BMT: 50mg/kg/day
  Other Names: Cytoxan
Drug: Mesna — Days 3 & 4 after BMT: 40 mg/kg IV
Drug: Sirolimus — Adjusted to maintain a serum trough level of 3-12 ng/mL, taken orally beginning on 5 days after BMT and taken to 1 year after BMT.
  Other Names: rapamycin, Rapamune®
Drug: Mycophenolate mofetil (MMF) — 15 mg/kg orally with maximum dose 3 mg/day beginning 5 days after BMT and taken to day 35 after BMT
Procedure: Bone marrow transplantation — Day 0 - Transplantation of hematopoietic cells derived from bone marrow of a donor to a recipient as treatment for hematologic disorders
Radiation: Total body irradiation — 200 cGy on the day before BMT. Radiation delivered to the entire body of the recipient to eradicate bone marrow cells in the recipient to prepare the recipient to receive the transplanted

SUMMARY:
Allogeneic blood or marrow transplantation (alloBMT) is a curative therapy for a variety of hematologic disorders, including sickle cell disease and thalassemia. Even when it is clear that alloBMT can give to these patients an improvement in their disease, myeloablative transplants have important toxicities and mortalities associated. The lack of suitable donors continues to be a limit to access to transplantation. Substantial progress has been made recently in the development of pre-treatment regimens that facilitate the sustained engraftment of donor marrow with reduced toxicity. Most of these regimens incorporate highly immunosuppressive drugs, which allow the reduction or elimination of myeloablative agents or total body irradiation without endangering the sustained engraftment of HLA-identical allogeneic stem cells. Preliminary results of non-myeloablative allogeneic stem cell transplantation suggest that the procedure can be performed in patients who are ineligible for myeloablative alloBMT, and that sustained remissions of several hematologic malignancies can be obtained.

ELIGIBILITY:
RECIPIENT INCLUSION CRITERIA

* Patients who are ineligible for BMT from an HLA-matched sibling donor can proceed to a haplo-BMT. Patients with an HLA-matched related donor will proceed to a matched BMT.
* Age 1-70 years
* Good performance status (ECOG 0 or 1; Karnofsky and Lansky 70-100)
* Patients and donors must be able to sign consent forms. First degree relative should be willing to donate
* Patients must be geographically accessible and willing to participate in all stages of treatment.
* Eligible diagnoses: Patients with sickle cell anemia such as sickle cell anemia (Hb SS), Hb Sβ° thalassemia, Hb Sβ+thalassemia, Hb SC disease, Hb SE disease, Hb SD disease, Hemoglobin SO- Arab disease HbS with hereditary persistence of fetal hemoglobin. Other significant hemoglobinopathies.

Plus one of the following:

* Attenuation of progressive disease (adults):
* Severe and debilitating vaso-occlusive pain despite hydroxyurea or regular blood transfusion therapy.
* Stroke and silent infarct; stroke or central nervous system event lasting more than 24 hours; MRI changes indicative of brain parenchyma damage and MRA evidence of cerebrovascular disease.
* Recurrent acute chest syndrome requiring exchange hospitalization.
* Chronic lung disease as defined by progressive restrictive disease irrespective of oxygen requirements.
* Chronic kidney disease, CKD stage II - IV
* Transfusion dépendent thalassemia

RECIPIENT EXCLUSION CRITERIA:

* Poor performance status (ECOG>1).
* Poor cardiac function: left ventricular ejection fraction<35%.
* Poor pulmonary function: FEV1 and FVC<40% predicted.
* Pulmonary hypertension moderate to severe by echocardiographic standards.
* Poor liver function: direct bilirubin >3.1 mg/dl
* HIV-positive
* Minor (donor anti-recipient) ABO incompatibility if an ABO compatible donor is available.
* Prior transfusions from donor or recipient if caused alloimmunization vs. donor cells.
* Women of childbearing potential who currently are pregnant (Beta-HCG+) or who are not practicing adequate contraception.
* Patients who have any debilitating medical or psychiatric illness that would preclude their giving informed consent or their receiving optimal treatment and follow-up. However, patients with history of stroke and significant cognitive deficit,that would preclude giving informed consent or assent will not be excluded, if they have a family member or significant other with Power of Attorney to also consent of their behalf.

CRITERIA FOR DONOR ELIGIBILITY:

* Weight ≥ 20kg and age ≥ 18 years or per institutional guidelines
* Donors must meet the selection criteria as defined by the Foundation for the Accreditation of Hematopoietic Cell Therapy (FAHCT) and will be screened per the American Association of Blood Banks (AABB). (AABB guidelines and the recipients will be informed of any deviations.)
* HLA-haploidentical first-degree relatives of the patient. Participants must be HLA typed at high resolution using DNA based typing at HLA-A, -B, -C and DRB1 and have available: An HLA haploidentical first degree relative donor (parents, siblings or half siblings, or children) with 2, 3, or 4 (out of 8) HLA-mismatches who is willing and able to donate bone marrow. A unidirectional mismatch in either the graft versus host or host versus graft direction is considered a mismatch. The donor and recipient must be HLA identical for at least one antigen (using high resolution DNA based typing) at the following genetic loci: HLA-A, HLA-B, HLA-C, and HLA-DRB1. Fulfillment of this criterion shall be considered sufficient evidence that the donor and recipient share one HLA haplotype, and typing of additional family members is not required.

When more than one donor is available, the donor with the lowest number of HLA allele mismatches will be chosen, unless there is HLA cross-match incompatibility or a medical reason to select otherwise, in which case donor selection is the responsibility of the PI, in consultation with the immunogenetics laboratory. In cases where there is more than one donor with the least degree of mismatch, donors will be selected based on the most favorable combination of:

* HLA compatibility in cross-match testing and
* ABO compatibility
* Donor age <40 years
* Avoid female donors for male recipients and
* Avoid CMV mismatched donor-recipient transplants:

HLA cross-matching (in order of priority):

* Mutually compatible (no cross-matching antibodies)
* Recipient non-cross-reactive with donor, donor cross-reactive with recipient
* Mutually cross-reactive

ABO compatibility (in order of priority):

* Compatible
* Major incompatibility
* Minor incompatibility
* Major and minor incompatibility
* Donors will be selected to minimize HLA mismatch in the Host-versus-graft direction.
* Donors fulfilling the following criteria are ineligible for registration onto this study:
* All donors will be screened by hemoglobin electrophoresis; donors with a clinically significant hemoglobinopathy are ineligible. Sickle trait is acceptable.

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2023-11 (Actual); Study Completion 2024-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Adetola A Kassim, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (3):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States
- Saint-Louis Hospital, Paris, France
- St Mary's Hospital, London, United Kingdom

REFERENCES:
- [Derived] Kassim AA, de la Fuente J, Nur E, Wilkerson KL, Alahmari AD, Seber A, Bonfim C, Simoes BP, Alzahrani M, Eckrich MJ, Horn B, Hanna R, Dhedin N, Rangarajan HG, Gouveia RV, Almohareb F, Aljurf M, Essa M, Alahmari B, Gatwood K, Connelly JA, Dovern E, Rodeghier M, DeBaun MR. An international learning collaborative phase 2 trial for haploidentical bone marrow transplant in sickle cell disease. Blood. 2024 Jun 20;143(25):2654-2665. doi: 10.1182/blood.2023023301. PMID 38493482
- [Derived] Aumann MA, Richerson W, Song AK, Davis LT, Pruthi S, Davis S, Patel NJ, Custer C, Kassim AA, DeBaun MR, Donahue MJ, Jordan LC. Cerebral hemodynamic changes after haploidentical hematopoietic stem cell transplant in adults with sickle cell disease. Blood Adv. 2024 Feb 13;8(3):608-619. doi: 10.1182/bloodadvances.2023010717. PMID 37883803
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-Myeloablative Conditioning and Bone Marrow Transplantation: Thymoglobulin: Day 9 before BMT: 0.5mg/kg IV; Days 8 & 7 before BMT: 2mg/kg IV
  Fludarabine: Days 6 and 2 before BMT: 30mg/m2/day IV
  Cyclophosphamide (CTX): Days 6 and 5 before BMT: 14.5mg/kg IV; Days 3 and 4 after BMT: 50mg/kg/day
  Mesna: Days 3 & 4 after BMT: 40 mg/kg IV
  Sirolimus: Adjusted to maintain a serum trough level of 3-12 ng/mL, taken orally beginning on 5 days after BMT and taken to 1 year after BMT.
  Mycophenolate mofetil (MMF): 15 mg/kg orally with maximum dose 3 mg/day beginning 5 days after BMT and taken to day 35 after BMT
  Bone marrow transplantation: Day 0 - Transplantation of hematopoietic cells derived from bone marrow of a donor to a recipient as treatment for hematologic disorders
  Total body irradiation: 200 cGy on the day before BMT. Radiation delivered to the entire body of the recipient to eradicate bone marrow cells in the recipient to prepare the recipient to receive the transplanted
Period: Overall Study
Arm/Group | Non-Myeloablative Conditioning and Bone Marrow Transplantation
Started | 26
Completed | 18
Not Completed | 8
Not completed — Lost to Follow-up | 4
Not completed — Not eligible | 1
Not completed — Failed engraftment | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Non-Myeloablative Conditioning and Bone Marrow Transplantation
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11
  Between 18 and 65 years | 15
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 22
  White | 1
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 21
  United Kingdom | 2
  France | 3

OUTCOME MEASURES:

1. Primary Outcome: Transplant-related Mortality (TRM)
Description: Defined as death in the absence of recurrent sickle cell disease or hemoglobinopathy
Time Frame: at 1 year after BMT
Population: participants in this study
Measure: Count of Participants; unit: Participants
Groups:
- Non-Myeloablative Conditioning and Bone Marrow Transplantation: Thymoglobulin: Day 9 before BMT: 0.5mg/kg IV; Days 8 & 7 before BMT: 2mg/kg IV
  Fludarabine: Days 6 and 2 before BMT: 30mg/m2/day IV
  Thiotepa: on Day -7 before BMT 10mg/kg (15 patients received this and one did not.)
  Cyclophosphamide: Days 6 and 5 before BMT: 14.5mg/kg IV; Days 3 and 4 after BMT: 50mg/kg/day
  Mesna: Days 3 & 4 after BMT: 40 mg/kg IV
  Sirolimus: Adjusted to maintain a serum trough level of 3-12 ng/mL, taken orally beginning on 5 days after BMT and taken to 1 year after BMT.
  Mycophenolate mofetil (MMF): 15 mg/kg orally with maximum dose 3 mg/day beginning 5 days after BMT and taken to day 35 after BMT
  Bone marrow transplantation: Day 0 - Transplantation of hematopoietic cells derived from bone marrow of a donor to a recipient as treatment for hematologic disorders
  Total body irradiation: 200 cGy on the day before BMT. Radiation delivered to the entire body of the recipient to eradicate bone marrow cells in the recipient to prepare the recipient to receive the transplanted
Arm/Group | Non-Myeloablative Conditioning and Bone Marrow Transplantation
Number analyzed (Participants) | 16
Participants | 0

2. Secondary Outcome: Number of Patients Who Developed Grade I-IV Acute Graft-vs.-Host Disease
Description: GVHD Severity was graded using the established National Institutes of Health's consensus criteria [36].
Time Frame: 2 years
Population: Participants in this study with median follow-up of 16.7 months (IQR, 6.5-30.8 months)
Measure: Count of Participants; unit: Participants
Groups:
- Non-Myeloablative Conditioning and Bone Marrow Transplantation: Thymoglobulin: Day 9 before BMT: 0.5mg/kg IV; Days 8 & 7 before BMT: 2mg/kg IV
  Fludarabine: Days 6 and 2 before BMT: 30mg/m2/day IV
  Thiotepa: on Day -7 before BMT 10mg/kg (15 patients received this and one did not.)
  Cyclophosphamide (CTX): Days 6 and 5 before BMT: 14.5mg/kg IV; Days 3 and 4 after BMT: 50mg/kg/day
  Mesna: Days 3 & 4 after BMT: 40 mg/kg IV
  Sirolimus: Adjusted to maintain a serum trough level of 3-12 ng/mL, taken orally beginning on 5 days after BMT and taken to 1 year after BMT.
  Mycophenolate mofetil (MMF): 15 mg/kg orally with maximum dose 3 mg/day beginning 5 days after BMT and taken to day 35 after BMT
  Bone marrow transplantation: Day 0 - Transplantation of hematopoietic cells derived from bone marrow of a donor to a recipient as treatment for hematologic disorders
  Total body irradiation: 200 cGy on the day before BMT. Radiation delivered to the entire body of the recipient to eradicate bone marrow cells in the recipient to prepare the recipient to receive the transplanted
Arm/Group | Non-Myeloablative Conditioning and Bone Marrow Transplantation
Number analyzed (Participants) | 16
Participants | 2

3. Secondary Outcome: Number of Patients With Donor Hematopoietic Chimerism in Peripheral Blood <95% at 6 Months After Mini-haploBMT
Description: Partially human leukocyte antigen (HLA)-mismatched bone marrow from first-degree relatives. Defined in percentages of donor cells in patient's peripheral blood, measured in 4 ways.
  * Mixed donor chimerism: > 0% but < 95%
  * Complete donor chimerism > 95%
  Any amount of donor chimerism after day 60 will be considered as having engrafted
Time Frame: Up to approximately 180 after mini-haploBMT
Population: Recipients of Haplo-BMT with PTCy and Thiotepa
Measure: Count of Participants; unit: Participants
Groups:
- Non-Myeloablative Conditioning and Bone Marrow Transplantation: Thymoglobulin: Day 9 before BMT: 0.5mg/kg IV; Days 8 & 7 before BMT: 2mg/kg IV
  Fludarabine: Days 6 and 2 before BMT: 30mg/m2/day IV Thiotepa: on Day -7 before BMT 10mg/kg
  Cyclophosphamide (CTX): Days 6 and 5 before BMT: 14.5mg/kg IV; Days 3 and 4 after BMT: 50mg/kg/day
  Mesna: Days 3 & 4 after BMT: 40 mg/kg IV
  Sirolimus: Adjusted to maintain a serum trough level of 3-12 ng/mL, taken orally beginning on 5 days after BMT and taken to 1 year after BMT.
  Mycophenolate mofetil (MMF): 15 mg/kg orally with maximum dose 3 mg/day beginning 5 days after BMT and taken to day 35 after BMT
  Bone marrow transplantation: Day 0 - Transplantation of hematopoietic cells derived from bone marrow of a donor to a recipient as treatment for hematologic disorders
  Total body irradiation: 200 cGy on the day before BMT. Radiation delivered to the entire body of the recipient to eradicate bone marrow cells in the recipient to prepare the recipient to receive the transplanted
Arm/Group | Non-Myeloablative Conditioning and Bone Marrow Transplantation
Number analyzed (Participants) | 15
Participants | 1

4. Secondary Outcome: Number of Participants With Hematologic and Non-hematologic Toxicities Following minihaploBMT
Description: Hematologic toxicity:
  -Absolute neutrophil count (ANC): consecutive values of < 500/µL on 3 different days after chemotherapy post-BMT Platelet count: consecutive values of < 20,000 µL on 3 different days after chemotherapy post-BMT
  Non-hematologic toxicities:
  -Toxicities necessitating hospitalization Toxicities grade 4 or above
  Meets the criteria of the following SAE:
  * Relapse of underlying disease
  * Grade 3 ocular toxicity not related to ocular GVHD
  * Grade 3 related non-hematologic toxicity
Time Frame: Day 60 after BMT
Population: Recipients of Haplo-BMT with PTCy and Thiotepa
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Myeloablative Conditioning and Bone Marrow Transplantation
Number analyzed (Participants) | 16
Participants
  Mucositis | 1
  Hepatic vessel clot | 1
  veno-occlusive disease of the liver | 1
  posterior reversible encephalopathy syndrome | 1
  Platelet refractory thrombocytopenis | 1
  Invasive fungal infection | 1
  Mycophenolate mofetilinduced gastritis | 1
  Duodenal ulcer-related gastrointestinal bleeding | 1
  Typhilitis | 1
  Encephalopathy | 1

ADVERSE EVENTS:
Time Frame: Day 100 after transplant
Arm/Group | Non-Myeloablative Conditioning and Bone Marrow Transplantation
All-Cause Mortality (participants affected / at risk) | 1/26
Serious Adverse Events (participants affected / at risk) | 9/26
Other Adverse Events (participants affected / at risk) | 0/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-Myeloablative Conditioning and Bone Marrow Transplantation (N=26)
Duodenal hemorrhage (Gastrointestinal disorders) | 1 (1)
Anaphylaxis (Nervous system disorders) | 1 (1)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 2 (2)
Fever (General disorders) | 2 (2)
Seizure (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Cognitive disturbancce (Nervous system disorders) | 1 (1)
Kidney injury (Renal and urinary disorders) | 2 (2)
Generalized weakness (General disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Epstein-Barr virus viremia (Infections and infestations) | 1 (1)
Hypotensive BSP (Vascular disorders) | 1 (1)
Febrile w/elevated WBC (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1)
Methicillin-resistant Staphylococcus aureus (MRSA) (Infections and infestations) | 1 (1)
Acute Graft-Versus-Host Disease (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-04): https://cdn.clinicaltrials.gov/large-docs/08/NCT01850108/Prot_SAP_000.pdf